CLINICAL TRIAL: NCT00073021
Title: A Double-Blind, Randomized, 6-Week, Parallel-Group Design Clinical Trial to Assess Safety and Efficacy of Asacol 4.8 g/Day (800 mg Tablet) Versus Asacol 2.4 g/Day (400 mg Tablet) for the Treatment of Moderately Active Ulcerative Colitis
Brief Title: Safety and Efficacy of Two Different Doses of Asacol in the Treatment of Moderately Active Ulcerative Colitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Warner Chilcott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2000082
Record Dates: First submitted 2003-11-13; First posted 2003-11-17 (Estimated); Results first posted 2011-07-28 (Estimated); Last update posted 2015-06-29 (Estimated); Status verified 2015-06

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Mesalamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Asacol 2.4 g/day (Active Comparator): Asacol (2.4 g/day)
  Interventions: Drug: Asacol 400 mg (mesalamine)
- Asacol 4.8 g/day (Experimental): Asacol (4.8 g/day)
  Interventions: Drug: Asacol 800 mg (mesalamine)

INTERVENTIONS:
Drug: Asacol 800 mg (mesalamine) — tablets, 4.8 g/day for 6 weeks, 2 - 800 mg Asacol tablets and 2 placebo tablets 3 times daily
  Arms: Asacol 4.8 g/day
Drug: Asacol 400 mg (mesalamine) — tablets, 2.4 g/day for 6 weeks, 2 - 400 mg Asacol tablets and 2 placebo tablets 3 times daily
  Arms: Asacol 2.4 g/day

SUMMARY:
This study is a prospective clinical study to evaluate the safety and efficacy of two different doses of Asacol for the treatment of moderately active ulcerative colitis. In addition, a new tablet formulation will be evaluated at one of the two doses.

ELIGIBILITY:
Inclusion Criteria:

* male or female between 18 and 75 years of age;
* have a confirmed diagnosis of ulcerative colitis with the extent varying from proctitis to pancolitis;
* currently demonstrating moderately active disease

Exclusion Criteria:

Patients will be excluded from admission to the study if they have/are:

* a history of allergy or hypersensitivity to salicylates or aminosalicylates;
* a history of extensive small bowel resection (>1/2 the length of the small intestine) causing short bowel syndrome;
* current renal or hepatic disease;
* participated in any drug or device clinical study within 30 days of entry;
* currently enrolled in any other clinical study;
* received any oral, intravenous, intramuscular, or rectally administered corticosteroids within 1 month prior to the Baseline Visit;
* received any other topical rectal therapy during the week prior to the Screening Visit;
* received immunomodulatory therapy including, but not limited to, 6-mercaptopurine, azathioprine, cyclosporine, or methotrexate within 3 months prior to the Baseline Visit;
* received a dose of mesalamine-containing compound by any route from which more than 1.6 g/day of mesalamine was available within 1 week prior to the Screening Visit (NOTE: 4 g/day of sulfasalazine and 4.5 g/day of balsalazide are equivalent to 1.6 g/day of mesalamine);
* received antibiotics, other than topical antibiotics, within 1 week prior to the Screening Visit;
* received aspirin (except for cardioprotective reasons up to a maximum dose of 325 mg/day) or NSAIDs within 1 week prior to the Baseline Visit;
* if female, positive pregnancy test, or lactating.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 386 (Actual)
Dates: Start 2000-09; Primary Completion 2003-09 (Actual); Study Completion 2003-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Krzeski, MD, Study Director — Procter and Gamble
Locations (57):
- United States (54):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - AGMG Clinical Research, Anaheim, California
  - Research Site, Los Angeles, California
  - Community Clinical Trials, Orange, California
  - AGMG Clinical Research, Orange, California
  - Research Site, Sacramento, California
  - Sharp Rees-Stealy Medical Group, San Diego, California
  - Research Site, Arvada, Colorado
  - Research Site, Englewood, Colorado
  - Center for Medical Research, LLC, Manchester, Connecticut
  - Center for GI Disorders, Hollywood, Florida
  - Research Site, Maitland, Florida
  - Advanced Gastroenterology Associates, Palm Harbor, Florida
  - Research Site, Zephyrhills, Florida
  - Southeast Research Associates, Marietta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - GI Research, Metairie, Louisiana
  - Louisiana Research Center, Shreveport, Louisiana
  - Digestive Disorders Associates, Annapolis, Maryland
  - Research Site, Baltimore, Maryland
  - Digestive Disease Associates, Baltimore, Maryland
  - Metropolitan Gastroenterology Group, Chevy Chase, Maryland
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - PharmaTrials, Inc., Hillsborough, New Jersey
  - Research Site, Forest Hills, New York
  - Long Island Clinical Research Associates, Great Neck, New York
  - Research Site, New York, New York
  - Carolinas Digestive Health Associates, Charlotte, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Statesville, North Carolina
  - Consultants for Clinical Research, Cincinnati, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - GI & Liver Consultants, Dayton, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Tulsa, Oklahoma
  - West Hills Gastroenterology Group, Portland, Oregon
  - Research Site, Altoona, Pennsylvania
  - Research Site, Hanover, Pennsylvania
  - Regional Research Institute, Jackson, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Houston Medical Research Associates, Houston, Texas
  - Research Site, Temple, Texas
  - Research Site, Ogden, Utah
  - Charlottesville Medical Research, Charlottesville, Virginia
  - Research Site, Fairfax, Virginia
  - Research Site, Fredericksburg, Virginia
  - Richmond GI Research, Richmond, Virginia
  - Research Site, Spokane, Washington
  - Wisconsin Center for Advanced Research, Milwaukee, Wisconsin
- Canada (2):
  - Research Site, Richmond, British Columbia
  - Research Site, Toronto, Ontario
- University of Puerto Rico, School of Medicine, San Juan, Puerto Rico

REFERENCES:
- [Derived] Orchard TR, van der Geest SA, Travis SP. Randomised clinical trial: early assessment after 2 weeks of high-dose mesalazine for moderately active ulcerative colitis - new light on a familiar question. Aliment Pharmacol Ther. 2011 May;33(9):1028-35. doi: 10.1111/j.1365-2036.2011.04620.x. Epub 2011 Mar 8. PMID 21385195
- [Derived] Lichtenstein GR, Ramsey D, Rubin DT. Randomised clinical trial: delayed-release oral mesalazine 4.8 g/day vs. 2.4 g/day in endoscopic mucosal healing--ASCEND I and II combined analysis. Aliment Pharmacol Ther. 2011 Mar;33(6):672-8. doi: 10.1111/j.1365-2036.2010.04575.x. Epub 2011 Jan 23. PMID 21255059

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began Feb. 28, 2001. Randomized 386 patients of which 117 had mild disease and 268 had moderate disease at baseline. Analysis only includes patients with moderate disease at baseline.
Groups:
- Asacol 2.4 g/Day: Two 400 mg Asacol tablets and 2 placebo tablets (matching 800 mg formulation) taken 3 times daily (morning, midday, evening).
- Asacol 4.8 g/Day: Two 800 mg Asacol tablets and 2 placebo tablets (matching 400 mg formulation) taken 3 times daily (morning, midday, evening).
Period: Overall Study
Arm/Group | Asacol 2.4 g/Day | Asacol 4.8 g/Day
Started | 139 (Subjects with Moderate Disease [PGA = 2] at Baseline) | 129 (Subjects with Moderate Disease [PGA = 2] at Baseline)
Completed | 113 | 113
Not Completed | 26 | 16
Not completed — Protocol Violation | 2 | 1
Not completed — Adverse Event | 4 | 4
Not completed — Withdrawal by Subject | 6 | 5
Not completed — Physician Decision | 3 | 1
Not completed — Lack of Efficacy | 11 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Asacol 2.4 g/Day | Asacol 4.8 g/Day | Total
Number analyzed (Participants) | 139 | 129 | 268
Age, Customized [Number; unit: Participants] — All Randomized Patients with Moderate Disease [PGA (Physician's Global Assessment) = 2] at Baseline
  Participants
    18 - 64 years | 126 | 118 | 244
    >= 65 years | 13 | 11 | 24
Sex: Female, Male [Count of Participants; unit: Participants] — All Randomized Patients with Moderate Disease [PGA = 2] at Baseline
  Participants
    Female | 77 | 75 | 152
    Male | 62 | 54 | 116
Race/Ethnicity, Customized [Number; unit: Participants] — All Randomized Patients with Moderate Disease [PGA = 2] at Baseline
  Participants
    Caucasian | 108 | 96 | 204
    Black or African American | 11 | 14 | 25
    Asian (Indian) | 1 | 2 | 3
    Asian (Oriental) | 1 | 3 | 4
    Hispanic | 16 | 11 | 27
    Multi-racial/other | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Treatment Success Patients at Week 6, ITT (Intent to Treat) Population
Description: Treatment success defined as complete response (PGA score 0 and complete resolution of stool frequency, rectal bleeding, PFA (patient's functional assessment), normal sigmoidoscopy) or partial response (improvement from baseline PGA and improvement in 1 clinical assessment [stool frequency, rectal bleeding, PFA, sigmoidoscopy] and no worsening in any other clinical assessments)
Time Frame: 6 Weeks
Population: ITT Population with Moderate Disease [PGA = 2] at Baseline
Measure: Number; unit: Percentage of Participants
Arm/Group | Asacol 2.4 g/Day | Asacol 4.8 g/Day
Number analyzed (Participants) | 130 | 124
Percentage of Participants | 59.2 | 71.8
Statistical Analysis 1: Comparison: Asacol 2.4 g/Day vs Asacol 4.8 g/Day; It was assumed that true rate of improvement for 2.4 g/day treatment group is 40% and for the 4.8 g/day group is 60%. To detect a true difference of 20% between these 2 groups with 2-sided test, type I error of 0.05 (alpha = 0.05), and power of 80%, 120 patients with moderately active ulcerative colitis were required per group to complete the study; Test type: Superiority or Other; p = 0.0357, Chi-squared; Difference in Success Rates = 12.543, 95% CI 2-sided [0.96 to 24.12]

2. Secondary Outcome: Change From Baseline in Ulcerative Colitis Disease Activity Index (UCDAI) at Week 6, ITT Population
Description: UCDAI - sum of clinical assessment scores (stool frequency score [0=normal, 1=1-2 stools > normal/day, 2=3-4 stools > normal/day, 3=5 or more stools > normal/day], rectal bleeding score [0=no blood seen, 1=streaks of blood with stool less than half of the time, 2=obvious blood with stool most of the time, 3=blood alone passed and PGA score [0=quiescent disease, 1=mild, 2=moderate, 3=severe]) and sigmoidoscopy score [0=normal, 1=mild, 2=moderate, 3=severe]
Time Frame: 6 weeks
Population: ITT Population with Moderate Disease [PGA = 2] at Baseline.
Measure: Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Asacol 2.4 g/Day | Asacol 4.8 g/Day
Number analyzed (Participants) | 130 | 124
Scores on a Scale | -3.2 (0.27) | -3.7 (0.27)
Statistical Analysis 1: Comparison: Asacol 2.4 g/Day vs Asacol 4.8 g/Day; Test type: Superiority or Other; p = 0.1594, ANOVA; Difference Between Means = -0.5, 95% CI 2-sided [-1.28 to 0.21]
Statistical Analysis 2: Comparison: Asacol 2.4 g/Day; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Compared to baseline; The 2-sample t-test will be used to examine the treatment effect
Statistical Analysis 3: Comparison: Asacol 4.8 g/Day; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Compared to baseline; Teh 2-sample t-test will be used to examine the treatment effect

3. Secondary Outcome: Percentage of Participants Whose Rectal Bleeding & Sigmoidoscopy Score Both Improved From Baseline to Week 6, ITT Population
Description: Rectal Bleeding - 0=no blood seen, 1=streaks of blood w/stool less than half of the time, 2=obvious blood w/stool most of the time, 3=blood alone passed Sigmoidoscopy Assessment Score - 0=normal (intact vascular pattern, no friability or granularity), 1=mild (erythema, diminished or absent vascular markings; mild granularity; friability), 2=moderate (marked erythema, granularity; absent vascular markings; bleeds with minimal trauma; no ulcerations) 3=severe (spontaneous bleeding, ulcerations)
Time Frame: 6 Weeks
Population: ITT Patients with Moderate Disease [PGA=2] at Baseline. Percentage of patients whose rectal bleeding AND sigmoidoscopy scores BOTH improved from baseline at Week 6
Measure: Number; unit: Percentage of Participants
Arm/Group | Asacol 2.4 g/Day | Asacol 4.8 g/Day
Number analyzed (Participants) | 130 | 124
Percentage of Participants | 59.8 | 63.6
Statistical Analysis 1: Comparison: Asacol 2.4 g/Day vs Asacol 4.8 g/Day; Test type: Superiority or Other; p = 0.5774, Chi-squared; Difference in Success Rates = 3.75, 95% CI 2-sided [-9.43 to 16.93]

4. Secondary Outcome: Percentage of Patients Whose Sigmoidoscopy Score Improved From Baseline to Week 6, ITT Population
Description: Sigmoidoscopy Assessment Score (0=normal intact vascular pattern, no friability or granularity, 1=mild erythema; diminished or absent vascular markings; mild granularity; friability, 2=moderate marked erythema, granularity; absent vascular markings; bleeds with minimal trauma; no ulcerations, 3=severe spontaneous bleeding, ulcerations)
Time Frame: 6 Weeks
Population: ITT Population with Moderate Disease [PGA=2] at Baseline
Measure: Number; unit: Percentage of Participants
Arm/Group | Asacol 2.4 g/Day | Asacol 4.8 g/Day
Number analyzed (Participants) | 130 | 124
Percentage of Participants | 69.0 | 75.2
Statistical Analysis 1: Comparison: Asacol 2.4 g/Day vs Asacol 4.8 g/Day; Test type: Superiority or Other; p = 0.2991, Chi-squared; Difference in Success Rates = 6.19, 95% CI 2-sided [-5.47 to 17.86]

5. Secondary Outcome: Percentage of Patients With an Improvement in Stool Frequency, ITT Population, Week 6
Description: 0=Normal stool frequency per day, 1=1-2 stools greater than normal per day, 2=3-4 stools greater than normal per day, 3=5 or more stools greater than normal per day
Time Frame: 6 Weeks
Population: ITT Patients with Moderate Disease [PGA=2] at Baseline
Measure: Number; unit: Percentage of Participants
Arm/Group | Asacol 2.4 g/Day | Asacol 4.8 g/Day
Number analyzed (Participants) | 130 | 124
Percentage of Participants | 71.3 | 74.0
Statistical Analysis 1: Comparison: Asacol 2.4 g/Day vs Asacol 4.8 g/Day; Test type: Superiority or Other; p = 0.6543, Chi-squared; Difference in Success Rates = 2.74, 95% CI 2-sided [-9.25 to 14.73]

6. Secondary Outcome: Percentage of Patients With Improvement in Rectal Bleeding, ITT Population, Week 6
Description: Rectal Bleeding (0=no blood seen, 1=streaks of blood with stool less than half of the time, 2=obvious blood with stool most of the time, 3=blood alone passed)
Time Frame: 6 Weeks
Population: ITT Population with Moderate Disease [PGA=2] at Baseline
Measure: Number; unit: Percentage of Participants
Arm/Group | Asacol 2.4 g/Day | Asacol 4.8 g/Day
Number analyzed (Participants) | 130 | 124
Percentage of Participants | 77.5 | 78.5
Statistical Analysis 1: Comparison: Asacol 2.4 g/Day vs Asacol 4.8 g/Day; Test type: Superiority or Other; p = 0.8542, Chi-squared; Difference in Success Rates = 1.05, 95% CI 2-sided [-10.19 to 12.29]

7. Secondary Outcome: Percentage of Patients With Improvement in Patient's Functional Assessment (PFA), ITT Population, Week 6
Description: PFA - 0=generally well, 1=fair, 2=poor, 3=terrible
Time Frame: 6 Weeks
Population: ITT Population with Moderate Disease [PGA=2] at Baseline
Measure: Number; unit: Percentage of Participants
Arm/Group | Asacol 2.4 g/Day | Asacol 4.8 g/Day
Number analyzed (Participants) | 130 | 124
Percentage of Participants | 70.5 | 69.6
Statistical Analysis 1: Comparison: Asacol 2.4 g/Day vs Asacol 4.8 g/Day; Test type: Superiority or Other; p = 0.8859, Chi-squared; Difference in Success Rates = -0.96, 95% CI 2-sided [-14.09 to 12.17]

8. Secondary Outcome: Percentage of Patients With Improvement in Physician Global Assessment (PGA)Score, ITT Population, Week 6
Description: PGA -Physician's Global Assessment - 0=quiescent disease (all parameters 0), 1=mild disease (parameters mostly 1's) 2=moderate (parameters mostly 2's), 3=severe (parameters mostly 3's) [parameters: combination of stool frequency, rectal bleeding, PFA & sigmoidoscopy findings] If scoring equal default to physician judgement.
Time Frame: 6 Weeks
Population: ITT Population with Moderate Disease [PGA=2] at Baseline
Measure: Number; unit: Percentage of Participants
Arm/Group | Asacol 2.4 g/Day | Asacol 4.8 g/Day
Number analyzed (Participants) | 130 | 124
Percentage of Participants | 73.5 | 83.2
Statistical Analysis 1: Comparison: Asacol 2.4 g/Day vs Asacol 4.8 g/Day; Test type: Superiority or Other; p = 0.0758, Chi-squared; Difference in Success Rates = 9.73, 95% CI 2-sided [-0.94 to 20.40]

9. Secondary Outcome: Mean Change From Baseline in Total Inflammatory Bowel Disease Questionnaire (IBDQ) at Week 3, All Randomized Patients
Description: IBDQ-32 questions divided into 4 categories: bowel, systemic, emotional and social. Each question graded with the following responses: 1-more than ever before, 2-extremely frequently, 3-very frequently, 4-moderate increase in frequency, 5-some increase in frequency, 6-slight increase in frequency or 7-not at all/normal; 1/worst thru 7/best. Scoring 32 - 224 - higher score better.
Time Frame: 3 Weeks
Population: All Randomized Patients with Moderate Disease[PGA=2] at Baseline. Questionnaire analyzable if patient answered 28 of 32 for total, 8/10 for bowel, 3/5 for systemic, 10/12 for emotional, 3/5 for social.
Measure: Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Asacol 2.4 g/Day | Asacol 4.8 g/Day
Number analyzed (Participants) | 139 | 129
Scores on a Scale | 30.4 (2.84) | 29.8 (2.60)
Statistical Analysis 1: Comparison: Asacol 2.4 g/Day vs Asacol 4.8 g/Day; Test type: Superiority or Other; p = 0.8308, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Asacol 2.4 g/Day; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Compared to baseline
Statistical Analysis 3: Comparison: Asacol 4.8 g/Day; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Compared to baseline

10. Secondary Outcome: Mean Change From Baseline in Total Inflammatory Bowel Disease Questionnaire (IBDQ) at Week 6, All Randomized Patients
Description: IBDQ-32 questions divided into 4 categories: bowel, systemic, emotional and social. Each question graded with the following responses: 1-more than ever before, 2-extremely frequently, 3-very frequently, 4-moderate increase in frequency, 5-some increase in frequency, 6-slight increase in frequency or 7-not at all/normal; 1/worst thru 7/best. Scoring 32-224 - higher score better.
Time Frame: 6 Weeks
Population: All Randomized Patients with Moderate Disease [PGA=2] at Baseline. Questionnaire analyzable if patient answered 28 of 32 for total, 8/10 for bowel, 3/5 for systemic, 10/12 for emotional, 3/5 for social.
Measure: Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Asacol 2.4 g/Day | Asacol 4.8 g/Day
Number analyzed (Participants) | 139 | 129
Scores on a Scale | 43.1 (3.5) | 40.4 (3.08)
Statistical Analysis 1: Comparison: Asacol 2.4 g/Day vs Asacol 4.8 g/Day; Test type: Superiority or Other; p = 0.5340, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Asacol 2.4 g/Day; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Compared to baseline
Statistical Analysis 3: Comparison: Asacol 4.8 g/Day; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Compared to baseline

11. Secondary Outcome: Percentage of Patients With Moderate, Left-Sided Disease at Baseline Classified as Treatment Success at Week 6, All Randomized Patients
Description: as for outcome 1
Time Frame: 6 Weeks
Population: All Randomized Patients with Moderate Disease [PGA=2] at Baseline. Left Sided Disease = proctitis, proctosigmoiditis or left-sided colitis
Measure: Number; unit: Percentage of Participants
Arm/Group | Asacol 2.4 g/Day | Asacol 4.8 g/Day
Number analyzed (Participants) | 105 | 97
Percentage of Participants | 60.0 | 71.1
Statistical Analysis 1: Comparison: Asacol 2.4 g/Day vs Asacol 4.8 g/Day; Test type: Superiority or Other; p = 0.0966, Chi-squared; Difference in Success Rates = 11.1, 95% CI 2-sided [-1.87 to 24.14]

12. Secondary Outcome: Percentage of Treatment Success Patients at Week 3, ITT Population
Description: as for outcome 1
Time Frame: 3 Weeks
Population: ITT Patients with Moderate Disease [PGA = 2] at Baseline
Measure: Number; unit: Percentage of Participants
Arm/Group | Asacol 2.4 g/Day | Asacol 4.8 g/Day
Number analyzed (Participants) | 130 | 124
Percentage of Participants | 51.5 | 61.3
Statistical Analysis 1: Comparison: Asacol 2.4 g/Day vs Asacol 4.8 g/Day; Test type: Superiority or Other; p = 0.1173, Chi-squared; Difference in Success Rates = 9.75, 95% CI 2-sided [-2.39 to 21.89]

ADVERSE EVENTS:
Time Frame: 6 week treatment period for each subject, February 28, 2001 thru April 15 2004
Arm/Group | Asacol 2.4 g/Day | Asacol 4.8 g/Day
Serious Adverse Events (participants affected / at risk) | 4/139 | 1/129
Other Adverse Events (participants affected / at risk) | 72/195 | 81/191
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Asacol 2.4 g/Day (N=139) | Asacol 4.8 g/Day (N=129)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Increased Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Cramping (Gastrointestinal disorders) | 1 (1) | 0 (0)
Exacerbation of Ulcerative Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Shoulder/Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Asacol 2.4 g/Day (N=195) | Asacol 4.8 g/Day (N=191)
Headache (Nervous system disorders) | 15 | 16
Pain, Abdominal (Gastrointestinal disorders) | 11 | 7
Infection (Infections and infestations) | 5 | 9
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 7 | 1
Diarrhea (Gastrointestinal disorders) | 6 | 8
Nausea (Gastrointestinal disorders) | 5 | 5
Rectal Disorder (Gastrointestinal disorders) | 5 | 5
Dyspepsia (Gastrointestinal disorders) | 5 | 4
Flu Syndrome (Infections and infestations) | 5 | 4
Colitis Ulcer (Gastrointestinal disorders) | 3 | 5
Fever (General disorders) | 4 | 4
Flatulence (Gastrointestinal disorders) | 6 | 2
Asthenia (General disorders) | 3 | 4
Cough Increased (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Rash (Skin and subcutaneous tissue disorders) | 4 | 2
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less